CLINICAL TRIAL: NCT00811148
Title: Establishment of a UF Brain Tumor Tissue Bank: Florida Center for Brain Tumor Research
Brief Title: Florida Center for Brain Tumor Research
Acronym: FCBTR
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: FCBTR; OCR13767 (Other: OnCore)
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Brain Tumors
Keywords: Brain Neoplasms; Central Nervous System Diseases; Central Nervous System Neoplasms; Brain Diseases; Nervous System Neoplasms
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Diseases; Central Nervous System Neoplasms; Brain Diseases; Nervous System Neoplasms | interventions — Tissue Banks

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, medical information, cerebrospinal fluid, blood and answers to Quality of Life questionnaires will be stored and made available to researchers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tissue Bank: Collection of clinical data and tumor tissue removed during brain surgeries for future research.
  Interventions: Procedure: Tissue Bank

INTERVENTIONS:
Procedure: Tissue Bank — Collection of clinical data and tumor tissue.

SUMMARY:
The purpose of this research study is to collect and store brain tumor tissue samples for future research. The samples will become part of the University of Florida Brain Tumor Tissue Bank/Florida Center for Brain Tumor Research. The goal is to find improved treatments and cures for brain tumors.

DETAILED DESCRIPTION:
The mission of the Florida Center for Brain Tumor Research is to discover cures for brain tumors and develop innovative brain tumor treatment modalities by providing a central repository for brain tumor biopsies and clinical information from individuals throughout the state of Florida, improving brain tumor biomedical research programs within the state of Florida, facilitating funding opportunities, fostering collaboration with brain tumor research organizations and other institutions, and fostering improved technology transfer of brain tumor research findings into clinical trials and widespread public use.

The Florida Center for Brain Tumor Research will collect and store left-over tissue that is not needed for medical care or diagnosis in a tissue bank in the Evelyn F. and William L. McKnight Brain Institute at the University of Florida. Tissue, medical information, cerebrospinal fluid, blood and answers to Quality of Life questionnaires will be stored and made available to researchers. Although developed for Florida, tumor tissue from all other states would be accepted.

ELIGIBILITY:
Inclusion Criteria:

* Children and adults scheduled to undergo brain surgery to remove tumor tissue.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults scheduled to undergo brain surgery to remove tumor tissue.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2006-03; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Collect and maintain clinical data and tumor tissue removed during brain surgeries. | 10 Years

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Rahman, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No